CLINICAL TRIAL: NCT05431166
Title: Virtual Yoga for Social Isolation and Loneliness in Rural Veterans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: Study00023836
Record Dates: First submitted 2022-03-29; First posted 2022-06-24 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-08

CONDITIONS: Loneliness; Social Isolation
Keywords: Veterans
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Intervention Model Description: Wait list Control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Treatment Group (Experimental): 8 weeks of Yoga Classes during first 8 weeks of study
  Interventions: Behavioral: Virtual Yoga at First 8 weeks
- Waitlist Control (Active Comparator): 8 weeks of Yoga Classes during second 8 weeks of study
  Interventions: Behavioral: Virtual Yoga at Second 8 weeks

INTERVENTIONS:
Behavioral: Virtual Yoga at First 8 weeks — 1 hour per week of virtual yoga delivered by an active movement therapist at the VA during the first 8 weeks of the study
  Arms: Immediate Treatment Group
Behavioral: Virtual Yoga at Second 8 weeks — 1 hour per week of virtual yoga delivered by an active movement therapist at the VA during the second 8 weeks of the study
  Arms: Waitlist Control

SUMMARY:
The overarching goal of this project is to decrease social isolation and loneliness through increased awareness and uptake of virtual yoga group classes among rural Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in VA Healthcare
* Residential address associated with VA Portland Health Care System that is "rural" or "highly rural; except among Collaborative Aging Research using Technology (CART) participants
* Valid contact info (mailing address, email, and phone number)
* High speed Internet access
* Positive screen for loneliness (NIH Toolbox Loneliness Scale Score greater or equal to 13)

Exclusion Criteria:

* Any VA or non-VA yoga visit in the preceding 12 months
* Visually or hearing impaired, or any mobility limitation that would impact computer/mobile device use, without availability of appropriate assistive devices
* Cognitive impairment, upcoming medical procedures, or significant unstable medical and psychiatric conditions that may limit study participation

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
UCLA Loneliness Scale, Version 3 | 10 Weeks
  Loneliness, higher scores indicate greater loneliness

SECONDARY OUTCOMES:
NIH Toolbox Loneliness Scale | 10 Weeks
  Loneliness, higher scores indicate greater loneliness
Modified Duke Social Support Index, Social Interaction Subscale | 10 Weeks
  Social Interaction Subscale
Modified Duke Social Support Index, Social Interaction by Relationship Subscale | 10 Weeks
  Social Interaction by Relationship Subscale
Promis Social Roles and Activities | 10 Weeks
  Measure on ability to participate in social roles and activities
Promis Satisfaction with Social Roles and Activities | 10 Weeks
  Measure on satisfaction with social roles and activities
PHQ-9 | 10 Weeks
  Depression measure
PC-PTSD-5 | 10 Weeks
  Post Traumatic Stress Disorder Measure
NIH CoRonavIruS Health Impact Survey (CRISIS) | 10 Weeks
  Selected items from this measure
CSQ-8 | 10 Weeks
  Adaption of CSQ-8, a Satisfaction measure
Treatment Delivery | 10 Weeks
  Treatment Delivery (Veteran Assessed)
Treatment Fidelity Checklist | 10 Weeks
  Treatment Fidelity Checklist (Assessed by Provider
Attitudes Toward Yoga | 10 Weeks
  Survey items on familiarity with yoga, reasons for participation in yoga, and expectations regarding yoga.
Sociodemographic Characteristics | 10 Weeks
  Items on age, race/ethnicity, sex, gender, military background, household cohabitation status, zip code, employment status, education, household income, spirituality
PEG (Pain, Enjoyment, General Activity) Scale | 10 Weeks
  Assessing Pain Intensity and Interference
SF-12 | 10 Weeks
  Assesses pain

CONTACTS AND LOCATIONS:
Locations (1):
- VA Portland Health Care System, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Teo AR, Benton MC, Hooker ER, Zaccari B, Hidalgo NJ, Newell S, Tuepker A, Greaves DW, Nicosia FM. Effect of telehealth yoga on loneliness and social isolation among rural older adults: a randomized controlled trial. Aging Ment Health. 2025 May;29(5):824-832. doi: 10.1080/13607863.2024.2449126. Epub 2025 Jan 10. PMID 39791606